CLINICAL TRIAL: NCT06420973
Title: A Single-arm, Multicenter, Phase II Study of RC48 Plus Platinum With or Without Bevacizumab in the Treatment of HER-2 Expression Platinum-Sensitive Recurrent Ovarian Cancer
Brief Title: RC48 Treatment for Platinum Sensitive Recurrent Ovarian Cancer With HER2 Expression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Hong Zheng, M.D., Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCVDODIIR017
Record Dates: First submitted 2024-05-11; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Carcinoma; Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48+carboplatin±bevacizumab (Experimental): RC48 (2.5mg/kg iv on d1 , every 21d for 6 cycles) + Carboplatin (AUC5 iv on d1 every 21d for 6 cycles)±Bevacizumab (7.5-15mg/kg iv on d1 every 21d for 6 cycles) for treatment followed by RC48 (2.5mg/kg iv on d1 , every 21d for 8 cycles)±Bevacizumab (7.5-15mg/kg iv on d1 every 21d for progress ) maintenance therapy.
  Interventions: Drug: RC48+carboplatin±bevacizumab

INTERVENTIONS:
Drug: RC48+carboplatin±bevacizumab — RC48 (2.5mg/kg iv on d1 , every 21d for 6 cycles) + Carboplatin (AUC5 iv on d1 every 21d for 6 cycles)±Bevacizumab (7.5-15mg/kg iv on d1 every 21d for 6 cycles) for treatment followed by RC48 (2.5mg/kg iv on d1 , every 21d for 8 cycles)±Bevacizumab (7.5-15mg/kg iv on d1 every 21d for progress ) maintenance therapy.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and quality of life scores of patients with HER2-expressing platinum-sensitive recurrent epithelial ovarian cancer treated with the combination therapy regimen of RC48 plus platinum with or without bevacizumab.

DETAILED DESCRIPTION:
This study set up a safety introduction period, during which the first 6 subjects who were initially enrolled in the study will slowly undergo safety monitoring. Each patient received RC48 [2.5 mg/kg, Q3W]+carboplatin (AUC5 d1 q3w) ± bevacizumab(7.5-15mg/kg d1 q3w) treatment. The monitoring time window is within 28 days after receiving the study drug treatment for the first time. If ≥ 2 dose limited toxicity (DLT) cases were observed in the first 6 subjects, and after evaluation by the research team, it was found that the toxicity was related to treatment with RC48, the initial dose of RC48 treatment for subsequent enrolled patients was adjusted to 2.0mg/kg, Q3W.

Treatment period: RC48+carboplatin ± bevacizumab, repeated every three weeks for a total of 6 cycles； Maintenance period: RC48± bevacizumab (if combined with bevacizumab during the treatment period, maintain treatment with RC48 in combination with bevacizumab; if not used during the treatment period, maintain treatment with RC48 monotherapy). Maintenance duration: Until disease progression or intolerable toxicity occurs, the longest duration of RC48 is 6 months (8 cycles).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged from 18 to 75 years old;
* Pathology confirmed the diagnosis of primary epithelial ovarian/fallopian tube/peritoneal carcinoma;
* Previous treatment lines ≥1 and ≤4, first-line treatment may include maintenance therapy after complete clinical or pathological response;Previously not receiving targeted HER2 drug therapy (including monoclonal antibodies and ADC drugs)
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1 at trial entry;
* Disease must be measurable by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1);
* Estimated life expectancy of more than 3 months;
* Local laboratory confirmed HER2 expression: IHC 1+, 2+, or 3+; Subjects were able to provide samples of the primary or metastatic site of the tumor for HER2 detection（Paraffin blocks, paraffin embedded sections or fresh tissue sections ）
* Adequate haematological, hepatic and renal functions defined by the protocol;
* Negative blood pregnancy test at Screening for women of childbearing potential; Highly effective contraception for female subjects if the risk of conception exists;

Exclusion Criteria:

* The pathological type is non epithelial ovarian/fallopian tube/peritoneal cancer or metastatic ovarian cancer;
* The patient has ≥ grade 2 peripheral neuropathy;
* Patients with active bleeding or pathological conditions with high risk of bleeding, such as known hemorrhagic diseases, coagulation disorders, or tumors involving large blood vessels;
* Suffering from central nervous system metastasis and/or cancerous meningitis. Except for stable brain metastases; 5.The toxicity caused by previous anti-tumor treatments has not yet recovered to CTCAE (version 5.0) level 0-1 (excluding 2nd degree hair loss);
* Patients who require parenteral hydration or nutrition and have evidence of partial intestinal obstruction or perforation;
* Except for patients with primary endometrial cancer or a history of primary endometrial cancer, unless all of the following conditions are met: stage not greater than I-B stage; No more than superficial muscle infiltration, no vascular or lymphatic infiltration; No poorly differentiated subtypes, including papillary fluid, clear cells, or other FIGO grade 3 lesions;
* For patients undergoing cell reduction surgery before treatment, if combined with bevacizumab, they must wait for at least 28 days before starting the treatment with bevacizumab;
* Have undergone major surgery within 4 weeks prior to the start of study administration and have not fully recovered;
* A large amount of pleural or ascitic fluid accompanied by clinical symptoms or requiring symptomatic treatment;
* Within 30 days of initial medication or expected to receive attenuated live vaccines during the study period;
* Serious arterial/venous thrombotic events or cardiovascular and cerebrovascular accidents that occurred within one year prior to drug administration were studied;
* There are systemic diseases that have not been controlled stably according to the judgment of the researcher, including diabetes, liver cirrhosis (Child Pugh Class B or C), interstitial pneumonia, obstructive pulmonary disease, etc;
* Clinically significant cardiovascular disease patients(According to the specific requirements of the plan);
* Individuals with active autoimmune diseases or immunodeficiency, or a history of the aforementioned conditions, including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, rheumatoid arthritis, inflammatory bowel disease, pituitary inflammation, vasculitis, nephritis, etc., shall not be included. The following exceptions apply: Patients with a history of autoimmune hypothyroidism who have received thyroid hormone replacement therapy may be included in the study. Patients with type 1 diabetes whose blood sugar can be controlled after treatment with insulin administration scheme can participate in this study;
* Subjects with a history of other malignant tumors within five years (excluding complete treatment for in situ cervical cancer, basal cell carcinoma, or squamous cell carcinoma skin cancer);
* Patients with congenital or acquired immune deficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 2000 IU / ml), hepatitis C (HCV antibody positive and HCV-RNA higher than the detection limit of the analytical method), or co infection of hepatitis B and hepatitis C;
* Severe infection (e.g. need for intravenous antibiotics, antifungal or antiviral drugs) occurred within 4 weeks before the first administration, or fever (>38.5%) of unknown reason occurred during the screening period/before the first administration；
* Currently participating in intervention clinical research treatment, or receiving other investigational drugs or research instruments within 4 weeks prior to the first administration; Not fully recovered from toxicity and/or complications caused by any intervention measures prior to initial administration (i.e. ≤ level 1 or reaching baseline, excluding fatigue or hair loss);
* Has a clear history of allergies and may have potential allergies or intolerance to the investigational drug and its similar biological agents;
* Individuals with a history of abuse of psychotropic substances who are unable to quit or have mental disorders;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-05-16 (Estimated); Primary Completion 2027-05-17 (Estimated); Study Completion 2027-09-17 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 2 years
  PFS is defined as time (in months) from date of randomization to the date of the first documentation of objective progressive disease (PD) or death due to any cause in the absence of documented PD (whichever occurs first). PFS will be determined according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) based on investigator response assessment.

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | Up to approximately 2 years
  ORR is defined as Investigator-assessed CR + PR, per RECIST 1.1
Disease Control Rate (DCR) | Up to approximately 2 years
  DCR is defined as the percentage of cases with remission (PR+CR) and stable disease (SD) after treatment in the evaluable cases.
Overall Survival（OS） | Up to approximately 2 years
  OS is defined as the time (in months) from randomization to the date of death, regardless of the actual cause of the subject's death.
Number of Participants With Adverse Events (AEs) | Up to approximately 2 years
  Assessment of the toxicity profile of regimen according to the National Cancer Institute Common Toxicity Criteria version 5.0 (NCI CTCAE v 5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Zheng, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No